CLINICAL TRIAL: NCT01222273
Title: Open-label Vitamin D Trial for Patients With Cystic Fibrosis and Allergic Bronchopulmonary Aspergillosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Joseph Pilewski, Associate Professor of Pediatrics, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO09090370; 7P50HL084932-04 (NIH)
Record Dates: First submitted 2010-10-14; First posted 2010-10-18 (Estimated); Results first posted 2018-03-29 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Cystic Fibrosis; Allergic Bronchopulmonary Aspergillosis
Keywords: cystic fibrosis; Allergic bronchopulmonary aspergillosis; A. fumigatus; Immune response
MeSH Terms: conditions — Cystic Fibrosis; Aspergillosis, Allergic Bronchopulmonary | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open label (Other): open label Vitamin D
  Interventions: Dietary Supplement: cholecalciferol (Vitamin D3)

INTERVENTIONS:
Dietary Supplement: cholecalciferol (Vitamin D3) — 4,000 IU of cholecalciferol (Vitamin D3) orally every day for six months
  Other Names: cholecalciferol

SUMMARY:
The purpose of this study is to see if giving people with CF and ABPA enough vitamin D to make their blood levels of the vitamin higher, will reduce the allergic response in their body and make the symptoms caused by ABPA better.

DETAILED DESCRIPTION:
Many patients with cystic fibrosis (CF) cough up mucus or have throat cultures that grow a common fungus called Aspergillus. In patients with CF, aspergillus is not known to cause direct damage to the lungs, but some patients respond with an allergic reaction that causes them to wheeze, cough, or have difficulty breathing. This allergic reaction is called ABPA. Current treatment for ABPA includes high dose steroids and an "anti-fungal" medicine. Treatment with steroids may be problematic for some people due to its side effects on blood sugar levels and the bones. Steroids are medications that decrease inflammation, including prednisone, medrol, dexamethasone and others.

Ongoing research at UPMC on the study "Mechanisms of Immune Tolerance in ABPA" has studied people with CF and ABPA versus those patients with CF that just grow A. fumigatus (Af) in the sputum, but do not have ABPA. You may have participated in this study. This study has shown that people with CF with the fungus, Af, in their sputum but who do not have ABPA have more of a certain type of cell in their blood that helps the body to regulate or suppress allergic reactions than those people with CF and ABPA.

Recent studies have demonstrated that Vitamin D is a critical factor in the development of these cells that suppress allergic reactions. People with CF, due to their pancreatic insufficiency that causes them to have difficulty absorbing fat, also have lower levels of the fat soluble vitamins which include vitamin D. In the study done at UPMC, "Mechanisms of Immune Tolerance in ABPA", people with CF and ABPA had significantly lower vitamin D levels than people with CF who did not have ABPA.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 12 years of age at enrollment
2. Confirmed diagnosis of CF based on the following criteria:

   1. One or more clinical features consistent with the CF phenotype AND (b or c)
   2. Positive sweat chloride > 60 mEq/liter (by pilocarpine iontophoresis)
   3. two identifiable mutations consistent with CF
3. Written informed consent (and assent when applicable) obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study.
4. Clinically stable at enrollment as assessed by the site investigator
5. Past or present respiratory culture positive for Aspergillus fumigatus
6. IgE ≥ 250 and/or presence of class II or higher aspergillus specific IgE on enrollment
7. Ability to comply with medication use, study visits and study procedures as judged by the site investigator -

Exclusion Criteria:

* 1. Systemic corticosteroids (1 mg/kg if < 20 kg or > 20 mg of prednisone per day),.

  2. Investigational drug use within 30 days of screening 3. Laboratory abnormalities at screening

  a. Serum Calcium > 11 mg/dl b. 25(OH) D > 50 ng/ml at screening. c. Creatinine ≥ 1.5, or estimated GFR <60 by Cockcroft-Gault or MDRD equation. d. LFT≥ 3xULN

  4. History of transplantation or currently on lung transplant list 5. Positive serum pregnancy test at screening (to be performed on all post-menarche females) 6. Pregnant, breastfeeding, or if post-menarche female, unwilling to practice birth control during participation in the study 7. Presence of a condition or abnormality that in the opinion of the site investigator would compromise the safety of the subject or the quality of the data 8. Diagnosis of HIV and a CD4+ T cell count below 500 cells/ml or active hepatitis B or C infection.

  9. Undergoing therapy for non-tuberculous mycobacterial infection

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph M Pilewski, MD, Principal Investigator — University of Pittsburgh; Jay K Kolls, MD, Study Director — University of Pittsburgh
Locations (2):
- United States (2):
  - Comprehensive Lung Center - Falk Clinic, Pittsburgh, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nguyen NL, Pilewski JM, Celedon JC, Mandalapu S, Blanchard ML, DeRicco A, Hartigan E, Alcorn JF, Kolls JK. Vitamin D supplementation decreases Aspergillus fumigatus specific Th2 responses in CF patients with aspergillus sensitization: a phase one open-label study. Asthma Res Pract. 2015;1:3. doi: 10.1186/s40733-015-0003-5. Epub 2015 Jun 4. PMID 27011794
- See also: Vitamin D supplementation decreases Aspergillus fumigatus specific Th2 responses in CF patients with aspergillus sensitization: a phase one open-label study — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4801182/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The CF Foundation patient registry will be queried for patients meeting inclusion/exclusion criteria. A recruitment letter will be sent to these patients. Additionally, patients/parents of patients will be approached regarding study participation by the investigator at routine clinic visits.
Groups:
- Cholecalciferol: 2000 Units of cholecalciferol once daily
  cholecalciferol (Vitamin D3): 4,000 IU of cholecalciferol (Vitamin D3) orally every day for six months
Period: Overall Study
Arm/Group | Cholecalciferol
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Subjects with CF with a prior history of clinically diagnosed ABPA
Arm/Group | Cholecalciferol
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.91 (2.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 7
BMI [Mean (Standard Deviation); unit: kg/m^2] | 22.5 (10.68)
IgE [Mean (Standard Deviation); unit: IU/mL] | 344.6 (284.9)
Asp IgE [Mean (Standard Deviation); unit: kUA/I] | 18.4 (14.7)
Genotype [Count of Participants; unit: Participants]
  ΔF508/R553X | 1
  ΔF508/612+ 1G-T | 1
  neg/ΔF508 | 1
  ΔF508/ΔF508 | 1
  MEG/G542X | 1
  ΔF508/1213delT | 1
  ΔF508/R1162X | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Aspergillus Induced IL-13 Responses in CD4+ T-cells
Description: To test the hypothesis that supplementation with Vitamin D in CF patients with ABPA will reduce Aspergillus induced IL-13 responses in peripheral CD4+ T-cells. Response confirmed for each individual patient and recorded as number of participants with response.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cholecalciferol
Number analyzed (Participants) | 7
Participants | 7

2. Secondary Outcome: Change in Patient Total IgE Levels
Description: To test the hypothesis that supplementation with Vitamin D in CF patients with ABPA will reduce total IgE levels by the end of the 24-week period
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Cholecalciferol
Number analyzed (Participants) | 7
IU/mL | 312.6 (77.66)

3. Secondary Outcome: Change in Patient Aspergillus Specific IgE Levels
Description: To test the hypothesis that supplementation with Vitamin D in CF patients with ABPA will reduce aspergillus specific IgE levels by the end of the 24-week period
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: kUA/I
Arm/Group | Cholecalciferol
Number analyzed (Participants) | 7
kUA/I | 11.73 (3.581)

ADVERSE EVENTS:
Time Frame: 6 months
Description: same as clinicaltrials.gov definitions
Arm/Group | Cholecalciferol
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes